CLINICAL TRIAL: NCT06721780
Title: AR Vs VR in Burns Dressing Changes
Acronym: AR vs VR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Buckinghamshire Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RXQ 1136
Record Dates: First submitted 2024-11-26; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-11

CONDITIONS: Burns Multiple

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Standard care (No Intervention): This is standard care (what they would normally receive if they were not enrolled into this study)
- Participants randomised to wear AR headset (Active Comparator): AR headset: MagicLeap 2 - running Divertini's "Watering Plants" world.
  Interventions: Device: Participants randomised to wear AR headset
- Participants randomised to wear VR headset (Active Comparator): VR Headset: Oculus Quest 2 - Running SyncVR's Relaxation and Pain control simulations
  Interventions: Device: Participants randomised to wear VR headset

INTERVENTIONS:
Device: Participants randomised to wear AR headset — Participants will use an AR headset that employs a distraction game specifically designed for children and young adults undergoing painful procedures.
  Arms: Participants randomised to wear AR headset
Device: Participants randomised to wear VR headset — Participants will utilise a VR headset, running a calming virtual environment or an interactive game during the dressing change.
  Arms: Participants randomised to wear VR headset

SUMMARY:
For children with burn injuries, changing their dressings can be one of the most traumatising experiences of their treatment journey. This process is not only distressing for the children but also for their parents and the healthcare professionals involved. Current methods to reduce this trauma include the use of play therapists, but such resources are often limited. There is good evidence that Augmented Reality (AR) and Virtual Reality (VR) can help by providing a distracting and immersive environment that eases pain and fear. However, no studies have yet compared these two modern technologies to see which is more effective

ELIGIBILITY:
Inclusion Criteria:

* • Participants presenting with guardians with parental responsibility, who are willing and able to consent to recruitment.

  * Aged 4-17 years
  * Presenting with burns requiring a dressing change, on their first attendance to the burns clinic.
  * Participating child is able to complete the FACES Pain Scale

Exclusion Criteria:

* • Children aged 4 or below

  * Those with severe cognitive impairment, visual disorders, facial burns or other conditions preventing the safe use of VR/AR technology.
  * Previous 'cybersickness' symptoms (nausea, dizziness).

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
determine the relative performance | 2 hours
  To determine the relative performance of AR and VR in pain and anxiety control during burns dressings changes in comparison to standard of care.
  Objective measures: Pulse rate, Respiratory rate

IPD SHARING:
Plan to Share IPD: No